CLINICAL TRIAL: NCT03869762
Title: A Phase II Study of Denosumab in Combination With Enzalutamide in Progressive Metastatic Castrate-resistant Prostate Cancer and Bone Metastases.
Brief Title: Denosumab in Combination With Enzalutamide in Progressive Metastatic Castrate-resistant Prostate Cancer and Bone Metastases.
Acronym: DICE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient accrual
Sponsor: Cancer Trials Ireland (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTRIAL-IE 17-17
Record Dates: First submitted 2019-03-08; First posted 2019-03-11 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Castration-resistant Prostate Cancer; Metastatic Cancer; Bone Metastases
Keywords: Castration-resistant; Progressive; Metastatic; Prostate Cancer; Bone Metastases
MeSH Terms: conditions — Neoplasm Metastasis; Prostatic Neoplasms | interventions — Denosumab; enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Denosumab & Enzalutamide (Experimental): 120mg subcutaneous injection on Day 1 of every four week cycle, for a maximum of 24 cycles, or until clinical disease progression, unacceptable toxicity, consent withdrawal or withdrawal for any other reason.
  160mg PO daily; (4 x 40 mg capsules) until confirmed clinical disease progression, unacceptable toxicity, consent withdrawal or withdrawal for any other reason)
  Interventions: Drug: Xgeva; Drug: Xtandi

INTERVENTIONS:
Drug: Xgeva — Denosumab is a human monoclonal antibody (IgG2) that targets and binds with high affinity and specificity to RANKL, preventing the RANKL/RANK interaction from occurring and resulting in reduced osteoclast numbers and function, thereby decreasing bone resorption and cancer induced bone destruction.
  Other Names: Denosumab
Drug: Xtandi — Enzalutamide is a potent androgen receptor signalling inhibitor that blocks several steps in the androgen receptor signalling pathway. Enzalutamide competitively inhibits binding of androgens to androgen receptors, inhibits nuclear translocation of activated receptors and inhibits the association of the activated androgen receptor with DNA even in the setting of androgen receptor overexpression and in prostate cancer cells resistant to anti-androgens.
  Enzalutamide treatment decreases the growth of prostate cancer cells and can induce cancer cell death and tumour regression.
  Other Names: Enzalutamide

SUMMARY:
Open-label phase II multi-centre single arm study of Denosumab in combination with enzalutamide in progressive metastatic castrate-resistant prostate cancer.

DETAILED DESCRIPTION:
This is an open-label phase II multi-centre single arm study of Denosumab in combination with enzalutamide in progressive metastatic castrate-resistant prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained prior to any study-related procedures.
2. Age ≥ 18 years and male.
3. ECOG performance status ≤ 2.
4. Histologically/cytologically confirmed adenocarcinoma of the prostate, and without neuroendocrine differentiation or small cell histology.
5. Documented metastatic disease with at least 1 bone metastasis on bone scan and confirmed, if necessary, by CT scan or MRI, if results of the bone scans are ambiguous. Patients with or without visceral involvement / lymph nodes (documented by RECIST 1.1) are allowed.
6. Patients must have documented Progressive disease (PD) either by radiographic or PSA criteria as defined in a) and b) below:

   1. For the Radiographic PD assessment, 2 sets of scans using the same imaging modality (ie CT/MRI or bone scan) and taken at separate time points are required to document radiographic disease progression during or following the patient's most recent anti-neoplastic therapy, (note: the 1st bone scan can be from before most recent therapy but the 2nd scan must show disease progression during or after the most recent therapy).

      For patients with bone disease, progression will be assessed following recommendations by the Prostate Cancer Working Group (PCWG3) (Appendix I): appearance of 2 or more new lesions on bone scan, confirmed, if necessary, by other imaging modalities (such as CT scan or MRI), if results of the bone scans are ambiguous).

      For patients with soft tissue lesions progression will be assessed using RECIST 1.1 criteria, (see Appendix C). Patients may have measurable or non-measurable disease according to RECIST criteria version 1.1 (see Appendix C)
   2. PSA progression as per PCWG3 (Appendix I) is defined as an increase in PSA, as determined by 2 separate measurements taken at least 1 week apart and confirmed by a third. If the third measurement is not greater than the second measurement, then a fourth measurement must be taken and must be greater than the second measurement for the patient to be eligible for the study. Furthermore, the confirmatory PSA measurement (i.e. the third or, if applicable, fourth PSA measurement) must be defined. If a patient has received prior anti-androgen therapy (e.g. bicalutamide), PSA progression must be evident and documented after discontinuation of anti-androgen therapy, (note: The 1st PSA reading taken to document disease progression when the patient presents can be while the patient is on Casodex or other ADT).
7. Prior surgical castration or concurrent use of an agent for medical castration (e.g. GnRH analogue) with testosterone at screening less than 1.73 nmol /l (50ng/dL).
8. Screening PSA ≥ 2 ng/mL.
9. Patients must agree to:

   * abstain from intercourse or
   * if the patient engages in sexual intercourse with a woman of childbearing potential, a condom and a highly effective birth control must be used (i.e. hormonal contraception associated with inhibition of ovulation, intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion or a vasectomy that has received medical assessment of the surgical success) during treatment and for 5 months after treatment.
10. Stable medical condition, including the absence of acute exacerbations of chronic illnesses, serious infections, or major surgery within 28 days prior to registration.
11. Life expectancy of 12 months or more based on general health and prostate cancer disease status as judged by the investigator.
12. Able to swallow study drug as whole tablet.
13. Adequate haematological, hepatic, and renal function.

    * Haemoglobin ≥ 10g/dL.
    * Neutrophils (ANC/AGC) ≥ 1500/mm³ (1.5 x 109/L).
    * Platelets ≥ (100 x 109/L).
    * Total bilirubin ≤ 1.5mg/dL (25.65 μmol/L) with the exception of Gilberts syndrome.
    * Both Alanine aminotransferase (ALT (SGPT)) and Aspartate aminotransferase (AST (SGOT) ≤ 3 x ULN with or without liver Metastasis.
    * Calculated creatinine clearance (CrCl) ≥ 30mL/min according to the Cockcroft and Gault formula (Appendix D).
    * Serum corrected Calcium within normal range and > 2 mmol/L
14. Continuous daily use of oral prednisone, oral dexamethasone, or other systemic corticosteroids is allowed prior to study entry but must be discontinued a minimum of 2 weeks prior to start of study treatment.

Exclusion Criteria:

1. Patients should not be receiving any other investigational agents for the treatment of prostate cancer or other diseases (within 30 days prior to registration).
2. Patients with GI tract disease resulting in an inability to take oral medication, malabsorption syndrome, a requirement for IV alimentation, prior surgical procedures affecting absorption, uncontrolled inflammatory GI disease (e.g., Crohn's disease, ulcerative colitis).
3. Have current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, or stable chronic liver disease per investigator assessment).
4. Prior therapy with orteronel, ketoconazole, aminoglutethimide, abiraterone or enzalutamide, denosumab or radium 223.
5. All anti-androgen therapy (including bicalutamide) is excluded within 6 weeks prior to first dose of study drug. Any other therapies for prostate cancer, other than GnRH analogue therapy, such as progesterone, medroxyprogesterone, progestins (megesterol), or 5-alpha reductase inhibitors (eg, finasteride or dutasteride), must be discontinued 2 weeks before the first dose of study drug. No prior bisphosphonates/Rank ligand inhibitors are allowed except when administered for bone density preservation in association with androgen deprivation therapy.
6. Prior chemotherapy for prostate cancer, with the exception of:

   * neoadjuvant/ adjuvant therapy as part of initial primary treatment for local disease that was completed 2 or more years prior to screening.
   * Patients who received prior docetaxol for castrate sensitive metastatic prostate cancer commencing with 120 days of ADT initation where total dose received did not exceed 450mg/m2
7. Diagnosis of or treatment for another systemic malignancy within 2 years before the first dose of study drug, or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with non-melanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
8. History of myocardial infarction, unstable symptomatic ischemic heart disease/ unstable angina, uncontrolled on-going arrhythmias of Grade >2 (National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5), pulmonary embolism, or any other cardiac condition (e.g. pericardial effusion restrictive cardiomyopathy) within 6 months prior to first dose of study drug. Patients with long QT, QTcF >470ms or uncontrolled hypertension are excluded.
9. New York Heart Association Class III or IV heart failure (see Appendix F).
10. History of seizure, underlying brain injury with loss of consciousness, stroke, transient ischaemic attack (TIA), cerebral vascular accident, primary brain tumours or brain metastases, brain arteriovenous malformation, alcoholism, or the use of concomitant medications that may lower the seizure threshold.
11. Known human immunodeficiency virus (HIV) infection, active chronic hepatitis B or C, life-threatening illness unrelated to cancer, or any ongoing serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with participation in this study. Patients will be tested for hepatitis B or C or HIV infection during screening if they are considered by the investigator to be at higher risk for these infections and have not been previously tested, or if testing is required by the independent ethics committee or institutional review board.
12. Prohibited medications, including drugs that are known to lower the seizure threshold or prolong QT interval are not permitted see section 7.4.2.
13. Patients with prior history of ONJ or osteomyelitis of the jaw, an active dental or jaw condition requiring oral surgery, non-healed dental/oral surgery, or any planned invasive dental procedure are excluded as confirmed by dental examination.
14. Patients with rare hereditary problems of fructose intolerance.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 7 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2019-01-12 (Actual); Study Completion 2019-01-12 (Actual)

PRIMARY OUTCOMES:
Radiographic progression free survival (rPFS) | 12 months
  Measured according to PCWG3 and RECIST 1.1 criteria. Result will be compared to historical rPFS in Enzalutamide be compared to historical rPFS in Enzalutamide

SECONDARY OUTCOMES:
Overall survival | 24 months
  Result will be compared to historical OS in Enzalutamide Enzalutamide
PSA progression free survival | 24 months
  Measured according to the PCWG3 criteria
Time to first skeletal-related event | 24 months
  Event will be calculated from the date of registration to the date of first skeletal-related event
Pain assessment | 24 Months
  Brief Pain Inventory - Short Form

CONTACTS AND LOCATIONS:
Overall Officials: Prof Ray McDermott, Principal Investigator — The Adelaide and Meath Hospital, Dublin, incorporating the National Children's Hospital
Locations (7):
- Ireland (7):
  - Galway University Hospital, Galway, Connacht
  - Sligo University Hospital, Sligo, Connacht
  - Adelaide and Meath incorporating National Children's Hopsital, Dublin, Leinster
  - St. Vincent's Hospital, Dublin, Leinster
  - Cork University Hospital, Cork, Munster
  - University Hospital Limerick, Limerick, Munster
  - University Hospital Waterford, Waterford, Munster